CLINICAL TRIAL: NCT03561701
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Oteseconazole (VT-1161) Oral Capsules in the Treatment of Subjects With Recurrent Vulvovaginal Candidiasis
Brief Title: A Study of Oral Oteseconazole (VT-1161) for the Treatment of Patients With Recurrent Vaginal Candidiasis (Yeast Infection)
Acronym: VIOLET
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mycovia Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VMT-VT-1161-CL-012
Record Dates: First submitted 2018-06-01; First posted 2018-06-19 (Actual); Results first posted 2021-12-20 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Recurrent Vulvovaginal Candidiasis
MeSH Terms: conditions — Candidiasis, Vulvovaginal | interventions — VT-1161

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oteseconazole (VT-1161) 150mg capsule (Experimental): Once daily for 7 days starting at Day 1, followed by once weekly for 11 weeks
  Interventions: Drug: Oteseconazole (VT-1161)
- Placebo capsule (Placebo Comparator): Once daily for 7 days starting at Day 1, followed by once weekly for 11 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oteseconazole (VT-1161) — Oteseconazole (VT-1161) 150mg capsule
  Arms: Oteseconazole (VT-1161) 150mg capsule
Drug: Placebo — matching placebo capsule
  Arms: Placebo capsule

SUMMARY:
Recurrent vulvovaginal candidiasis (RVVC), also known as recurrent yeast infections, is defined as at least 3 episodes of acute VVC in the past 12 months. Several properties of oteseconazole (VT-1161) suggest that it might be a safer and more effective treatment for RVVC than other oral antifungal medicines.

This study will evaluate the effectiveness and safety of oteseconazole (VT-1161) for the treatment of RVVC and consists of 2 parts. The first part of the study is a 2-week period for the treatment of the patient's current VVC episode with 3 150mg doses of fluconazole. The 2nd part consists of 12 weeks, when the patient will take either oteseconazole (VT-1161) 150 mg or a placebo (according to a random assignment), and then a 36-week follow-up period.

In addition, at participating sites, an amendment to the study allows US patients who complete the initial 48 weeks without experiencing a confirmed RVVC episode to continue in a 48-week observational extension period designed to evaluate the continued effectiveness of oteseconazole (VT-1161).

This study is identical to VMT-VT-1161-CL-011.

ELIGIBILITY:
Key Inclusion Criteria:

* 3 or more episodes of acute VVC in the past 12 months
* Positive KOH or Gram stain test
* Total vulvovaginal signs and symptoms score of ≥3 at screening visit
* Total vulvovaginal signs and symptoms score of <3 at baseline visit
* Must be able to swallow pills

Key Exclusion Criteria:

* Presence or a history of another vaginal or vulvar condition(s)
* Evidence of major organ system disease
* History of cervical cancer
* Poorly controlled diabetes mellitus
* Pregnant
* Recent use of topical or systemic antifungal or antibacterial drugs
* Recent use of immunosuppressive or systemic corticosteroid therapies

Min Age: 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2020-10-13 (Actual); Study Completion 2021-08-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - 31215, Phoenix, Arizona
  - 31227, Little Rock, Arkansas
  - 31217, Los Angeles, California
  - 31240, Hartford, Connecticut
  - 31204, Homestead, Florida
  - 31233, North Bay Village, Florida
  - 31255, Wichita, Kansas
  - 31245, Hagerstown, Maryland
  - 31223, Winston-Salem, North Carolina
  - 31244, Columbus, Ohio
  - 31229, Columbus, Ohio
  - 31222, Englewood, Ohio
  - 31218, Jackson, Tennessee
  - 31232, Frisco, Texas

REFERENCES:
- [Derived] Sobel JD, Donders G, Degenhardt T, Person K, Curelop S, Ghannoum M, Brand SR. Efficacy and Safety of Oteseconazole in Recurrent Vulvovaginal Candidiasis. NEJM Evid. 2022 Aug;1(8):EVIDoa2100055. doi: 10.1056/EVIDoa2100055. Epub 2022 Jul 26. PMID 38319878
- [Derived] Vanreppelen G, Nysten J, Baldewijns S, Sillen M, Donders G, Van Dijck P. Oteseconazole (VIVOJA) for prevention of recurrent vulvovaginal candidiasis. Trends Pharmacol Sci. 2023 Jan;44(1):64-65. doi: 10.1016/j.tips.2022.10.004. Epub 2022 Nov 14. No abstract available. PMID 36396498

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 425 subjects were enrolled in a 2-week Induction Phase after providing consent. During the Induction Phase, subjects received 3 sequential 150mg of fluconazole administered 72 hours apart. Subjects whose presenting acute VVC (vulvovaginal candidiasis) episode resolved during the Induction Phase (a total of 330) entered a 48-week Maintenance Phase comprised of a 12-week treatment period and a 36-week follow-up period.
Groups:
- Oteseconazole (VT-1161): 1 oteseconazole 150mg capsule once daily for 7 days starting at Day 1, then once weekly for 11 weeks
- Placebo: 1 placebo capsule once daily for 7 days starting at Day 1, then once weekly for 11 weeks
Period: Overall Study
Arm/Group | Oteseconazole (VT-1161) | Placebo
Started | 220 | 110
Completed | 191 | 91
Not Completed | 29 | 19

BASELINE CHARACTERISTICS:
Population: Four of the 330 subjects entering the 48-week Maintenance Phase were excluded from the ITT population. The numbers in the results sections reflect the ITT population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Oteseconazole (VT-1161) | Placebo | Total
Number analyzed (Participants) | 218 | 108 | 326
Age, Continuous [Median (Standard Deviation); unit: years] | 34 (9.4) | 36 (10.8) | 34 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 218 | 108 | 326
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 23 | 8 | 31
  White | 193 | 96 | 289
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  Belgium | 18 | 8 | 26
  Czechia | 51 | 22 | 73
  Hungary | 8 | 3 | 11
  Romania | 44 | 28 | 72
  Ukraine | 17 | 9 | 26
  United States | 80 | 38 | 118

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With 1 or More Culture-verified Acute VVC Episodes During the Maintenance Phase of the Study in the Intent-to-treat (ITT) Population.
Description: The primary efficacy outcome measure was the percentage of subjects with 1 or more culture-verified acute VVC episodes during the maintenance phase (post-randomization through Week 48) in the intent-to-treat population. An acute VVC episode during the maintenance phase (considered a recurrent episode) was defined as a positive fungal culture for Candida species and a clinical signs and symptoms score of ≥3. To calculate the signs and symptoms score, each vulvovaginal sign (erythema, edema, excoriation) and symptom (itching, burning, irritation) was scored using the following scale, with a higher score indicating a worse outcome.
  0 = none (complete absence of any sign or symptom), 1 = mild (slight), 2 = moderate (definitely present), 3 = severe (marked, intense)
Time Frame: Maintenance phase (post-randomization through Week 48)
Population: Analysis was performed on the ITT population which included all randomized subjects except the 4 excluded subjects. Missing values were imputed with multiple imputation using the following auxiliary information: region, treatment, baseline body mass index, baseline age, ethnicity, and visit.
Measure: Number; unit: percentage of subjects
Groups:
- Oteseconazole (VT-1161): 1 oteseconazole150mg capsule once daily for 7 days starting at Day 1, then once weekly for 11 weeks
Arm/Group | Oteseconazole (VT-1161) | Placebo
Number analyzed (Participants) | 218 | 108
percentage of subjects | 3.9 | 39.4

ADVERSE EVENTS:
Time Frame: Day 1 through Week 48 of the study
Description: The safety population was defined as all randomized subjects who received at least 1 dose of investigational product (3 subjects in the oteseconazole group did not receive investigational product). Treatment-emergent adverse events were defined as adverse events that occurred after the subject received her initial dose of investigational product.
Arm/Group | Oteseconazole (VT-1161) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/217 | 0/110
Serious Adverse Events (participants affected / at risk) | 7/217 | 5/110
Other Adverse Events (participants affected / at risk) | 112/217 | 63/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oteseconazole (VT-1161) (N=217) | Placebo (N=110)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Severe acute respiratory syndrome (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Motor dysfunction (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (4)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oteseconazole (VT-1161) (N=217) | Placebo (N=110)
Bacterial vaginosis (Infections and infestations) | 14 (23) | 6 (7)
Nasopharyngitis (Infections and infestations) | 11 (14) | 7 (9)
Urinary tract infection (Infections and infestations) | 12 (16) | 4 (6)
Influenza (Infections and infestations) | 6 (7) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 7 (7)
Cystitis (Infections and infestations) | 5 (6) | 3 (6)
Sinusitis (Infections and infestations) | 5 (7) | 2 (2)
Herpes simplex (Infections and infestations) | 0 (0) | 3 (3)
Tonsillitis (Infections and infestations) | 1 (1) | 2 (2)
Tooth infection (Infections and infestations) | 1 (1) | 2 (2)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 2 (5)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 2 (5)
Severe acute respiratory syndrome (Infections and infestations) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 18 (27) | 7 (7)
Migraine (Nervous system disorders) | 4 (7) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 4 (6) | 6 (8)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 3 (3) | 2 (2)
Dysmenorrhoea (Reproductive system and breast disorders) | 2 (2) | 2 (4)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 2 (3)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 6 (6) | 2 (2)
Vomiting (Gastrointestinal disorders) | 6 (6) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 2 (3)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Neither institution nor investigator can disclose information pertaining to study until sponsor issues multi-center publication. If multi-center publication is not issued within 18 months of study completion and database lock at all sites, sponsor has 30 days from receipt to review institution's and/or investigator's communication and can require removal of confidential information other than study data and/or delay release of institution's and/or investigator's communication for 60 days.

DOCUMENTS (2):
  • Study Protocol (2019-10-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT03561701/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-31): https://cdn.clinicaltrials.gov/large-docs/01/NCT03561701/SAP_001.pdf